CLINICAL TRIAL: NCT03413826
Title: Exercise and Weight Control: A Search for Biological and Neurobehavioral Compensatory Mechanisms That Defend Against Exercise-Induced Negative Energy Balance
Brief Title: Exercise and Weight Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kentucky (Other)
Responsible Party: Principal Investigator, Kyle Flack, Principle Investigator, University of Kentucky
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 17-0758-F2L
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Obesity; Exercise Reinforcement
Keywords: weight loss; exercise; reinforcement; compensation
MeSH Terms: conditions — Obesity; Weight Loss; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Baseline demographic and physical characteristics will be reported as means and standard errors. Baseline group (6 days/week, 2 days per week exercise, sedentary control) differences will be tested with one-way ANOVA. Alterations in accumulated negative energy balance, body composition, RRVfood, RRVexercise, dietary intake, energy expenditure, exercise discomfort, hunger/satiety hormones, and fitness will be tested with two-way repeated measures analysis of variance (RMANOVA) with group treated as a between-subjects variable and time treated as a within subjects variable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 6 Days per week (Experimental): This group will exercise 6 days per week and expend 3,000 kcal per week for 12 weeks
  Interventions: Behavioral: Exercise
- 2 Days per week (Experimental): This group will exercise 2 days per week and expend 3,000 kcal per week for 12 weeks
  Interventions: Behavioral: Exercise
- control (No Intervention): This group will remain sedentary for 12 weeks

INTERVENTIONS:
Behavioral: Exercise — The intervention groups will perform aerobic exercise for 12 weeks, expending 3,000 kcal of energy per week.
  Arms: 2 Days per week; 6 Days per week

SUMMARY:
The objective of this project is to determine the biological, neurobehavioral, and behavioral compensatory responses to exercise training-induced energy deficits in overweight to obese men and women. Participants will engage in exercise at either 2 days or 6 days per week for 12 weeks and have body composition assessed via DXA before and after the exercise intervention. Accumulated energy balance (weight loss converted to kcal) will be compared to exercise energy expenditure to determine each individual's level of compensation, termed compensation index. Predictors of compensation index that will be assessed will include hunger/satiety hormone concentrations at rest and in response to a meal, reward driven feeding, changes in metabolic rate, and energy intake throughout the intervention. Exercise reinforcement and physical activity will also be assessed as a separate aim to determine if exercise reinforcement can be increased and if this can promote greater habitual physical activity after the intervention has ceased.

DETAILED DESCRIPTION:
Study Design: A factorial design will be employed with exercise frequency (6 days/week or 2 days/week) treated as a between-subjects variable and time (baseline, end of training, end follow-up) treated as a within subjects variable. Subjects will be randomly assigned to exercise groups (6 days/week, 2 days/week) or sedentary control. The control group will be offered the intervention (personalized exercise plan, provided membership to YMCA) after follow-up measures.

Study Population:

This study will aim to complete all assessments on 60 participants

Inclusion Criteria:

* Male or female between the ages of 18 and 40
* Participants must be overweight to obese (BMI 25-35 kg/m2) Not pregnant or lactating or planning to become pregnant in the next 6 months
* No limitations to safely participating in physical activity

Exclusion Criteria:

* Currently dieting to lose weight and no weight loss or gain >2kg over the past 3 months,
* Taking any medications that affect energy expenditure or eating,
* Regularly exercising (planned and structured aerobic or resistance activity).
* Participants must have no major health problems, cannot have known cardiovascular (cardiac, peripheral vascular, cerebrovascular), pulmonary (COPD, interstitial lung disease, cystic fibrosis) or metabolic (diabetes, thyroid disorders, renal or liver disease) disease.
* Tobacco use
* Have a medical condition that prevents safe exercise.

Appropriateness of exercise will be screened using a Health History and Physical Activity Readiness Questionnaire. Subjects will taste and rate their liking of the study foods. Subjects must have a liking of at least 5 out of 10 for 50% of the study foods. Subjects will provide informed consent before participation. There are no hypotheses on gender or race effects and we will strive to recruit a representative sample that includes all gender and ethnic groups.

Specific hypotheses include:

H1: (Primary) Accumulated negative energy balance will be greater when exercising 2 times per week than exercising 6 times per week at 3000 kcal/week for 12 weeks.

H2: The RRVfood will increase more in response to 6 weekly exercise sessions than 2 sessions after 12 weeks of exercise.

H3: Energy intake will increase more in response to 6 weekly exercise sessions than 2 sessions after 12 weeks.

H4: Changes in GLP-1 concentration and RRVfood will be positively associated. H5: GLP-1, PYY, CCK, leptin, and pancreatic polypeptide concentrations will decrease in response to a meal more with 6 weekly exercise sessions than 2 sessions.

H6: Ghrelin concentrations will increase in response to a meal more with 6 weekly exercise sessions than 2 sessions.

H7: RRVexercise will increase more in response to 2 weekly exercise sessions than 6 sessions after 12 weeks.

H8: Tolerance to exercise discomfort will increase more in response to 2 weekly exercise sessions than 6 sessions after 12 weeks.

H9: The RRVexercise and tolerance to exercise discomfort will be positively associated with maintenance of exercise behaviors 4 weeks after the intervention (week 16).

H10: Changes in hunger hormones/peptides after 12 weeks of exercise will predict weight loss maintenance at week 17.

Research Procedures:

During the initial visit, participants will be informed about the study and have any questions answered. If deemed eligible and the participant desires to participate, they will be asked to provide written informed consent. After signing the consent, participants will fill out a demographic form, a medical history form and Physical Activity Readiness form, and be measured for anthropometrics (height and weight). These forms will be stored in a locked file cabinet in Dr. Flack's office separate from other study files. Subjects will also be provided an ActiGraph device to wear for the following week to monitor free-living physical activity and complete the Preference for and Tolerance of the Intensity of Exercise Questionnaire (PRETIE-Q), the Behavioral Regulation in Exercise Questionnaire (BREVQ-3), and the vendor form, so a payment can be processed) at this time.

Outcome visits: Outcome measures will be completed during baseline and immediately following the 12 weeks of training (Post/ week 13). Outcome measures will be completed at the CCTS, laboratory space in Funkhouser (room 117), Joe Craft Football Training Facility, or the Human Performance Laboratory as needed. The sequential order of the visits to measure outcomes is flexible in order to meet the scheduling complexities of participants.

Accelerometer administration: occurs at screening, after post-training assessments (week 14), and after follow-up assessments (week 19). Subjects will wear an accelerometer for seven consecutive days after receiving the accelerometer to measure usual physical activity. This will be scheduled so no exercise tests or sessions will fall on the 7 days wearing the monitor. This will be administered on participants' initial visit to Funkhouser 117 where they will also sign the consent form.

Surveys, taste test, height, weight: Will occur at screening, post-training/week 13, and follow up/week 18. The taste test will be used to determine the foods to be used in the RRVfood test. This visit will occur in Funkhouser 117.

RRVfood test: Will occur at weeks -1 or -2, 13, and 18. Subjects will report 2 to 3 hours postprandial to room 117 Funkhouser and complete a task where they will earn points towards their chosen foods.

RRVexercise test: Will occur at weeks -2 or -3, 13, and 18 at the Human Performance Laboratory (MDS, B04). subjects will sample for 2 minutes each and rate their liking of the 3 exercise options (treadmill, elliptical ergometer, or cycle ergometer) and sedentary alternatives (magazines, puzzles, card games). This testing can take place in the morning or afternoon, but will occur at the same time of day for a given subject.

BodPod + RMR test: Will occur at weeks -1 or -2, and 13. Subjects will report at least 10 hours postprandial and be assessed for their body composition (BodPod) and resting metabolic rate (RMR) at Funkhouser 117.

CCTS Meal test visit Will occur at weeks -1 or -2, and 13. Subjects will arrive to the CCTS (Center for Clinical and Transnational Science) on the UK campus at least 10 hours postprandial and have an IV-catheter placed and fasted blood sample collected. Subjects will then be administered a standardized breakfast and have blood drawn immediately after breakfast (-2.75), and every 15 minutes during the first hour (-2.5, -2.25, -2 hr) and then every 30 minutes thereafter (-1.5, -1, -0.5, 0) for a total testing time of 3 hrs. Subjects will also complete VAS scales for hunger and satiety at each blood draw time point.

CCTS Exercise test and DXA visit Will occur at weeks -1 or -2, week 6, week 13 Participants will report to the CCTS to perform a graded exercise test to determine kcal expended per minute at different heart rate intensities using indirect calorimetry. This information will be used to set the intensity and duration of their exercise training sessions during the intervention period of the study. This will be performed at baseline, on weeks 6 - 7, and after training. The mid-point measure will be used to adjust the duration and intensity of the exercise training sessions to account for any improvements in aerobic fitness. The post-time point measure will be used to determine aerobic fitness improvements. Prior to this test participants will also have a DXA scan preformed.

Additional DEXA test: Will occur at weeks -1 or -2 and 13. Subjects will report to the Joe Craft Football Training Facility to have an additional DXA performed on the UK athletics' Norland model DXA, a different model than the "gold standard" iDXA used at the CCTS.

Food Diary: for weeks -3, 4, 8, 12, 17 participants will record all foods they eat with details on quantity and cooking methods in a dietary intake record.

Exercise session download meeting: Once per week during the exercise intervention (weeks 1-12) participants will return to Funkhouser 117 to have their exercise sessions for the previous week downloaded to ensure compliance.

Intervention: For the exercise treatments, participants will engage in aerobic exercise (treadmill, stationary bike, elliptical) to induce a 3000 kcal/week energy expenditure exercising either 6 sessions per week (500 kcal per session) or 2 sessions per week (1500 kcal per session). The exercise intervention will last 12 weeks, followed by one week of post-testing and an unsupervised 4-week period where participants may exercise or not before final follow-up assessments at week 17. Exercise will occur at a moderate to difficult intensity and prescribed based on individual rates of energy expenditure (kcal/min) at different heart rate zones. Most exercise will occur at 65% of HRR, an intensity commonly prescribed for sedentary individuals beginning an exercise program [28]. The 6 session per week group should be able to complete the session in 20 to 60 min, while the 2 session per week group may take between 1.5 and 2.5 hours based on how many calories subjects burn exercising at 65% HHR. Subjects can take rest breaks as necessary during the exercise sessions. The first 2 to 5 exercise sessions will be supervised by research staff to introduce subjects to the use of the equipment and to ensure participants will be able to exercise for the prescribed time to meet their energy-expenditure goal. Then, exercise sessions will be supervised on an as needed basis in order to encourage compliance. To verify treatment implementation, subjects will wear a chest-strap heart rate monitor. Missed sessions (unless due to injury or illness) will be compensated for during the following sessions or made-up on another day. Heart rate and workout data will be reviewed by the research staff every week. Subjects will be able to use a 12-week pass to the Lexington-area YMCA(s) to assure access to exercise facilities if needed.

Measurements

Height and Weight. Body weight will be measured with a Tanita bioelectrical impedance scale after voiding. Subjects will wear scrubs or shorts and a t-shirt and no shoes when being weighed. Height will be with a stadiometer and standard anthropometric technique. These measurements will occur at screening to determine if subjects meets BMI inclusion criteria.

Food reinforcement task. Subjects will report 2-4 hr post-prandial to Funkhouser 117. RRVfood is assessed by evaluating the number of responses (mouse button presses) a participant is willing to complete to gain access to food. The foods used in the task were chosen to allow subjects to choose foods that are often considered both "junk" foods and "healthy" snacks with similar nutrient densities. The experimental environment will include two personal computers on separate workstations. At one station is the computer on which the participant can earn points towards their most liked junk food, with the other station being set up for them to earn points for their most liked healthy food. The most liked foods of each category are determined at screening by tasting a small portion of each food and rating each using a Likert-type scale. Participants can freely go back and forth between stations. The program used for the reinforcement task presents a game that mimics a slot machine. A point is earned each time the 3 shapes that appear with each mouse button press match in shape and color. Access to the alternatives is dependent on earning points, which can be exchanged for access to the reinforcers. For every 5 points earned, the subject will receive a 70-100 kcal portion of the food they were working for. Points are delivered on independent progressive fixed-ratio schedules. The schedules of reinforcement for food and reading begin at a fixed ratio of 4 and then doubles (8, 16, 32, […] 2048) each time 5 points are earned. For instance, the participant initially has to click the mouse four times to earn each point, but after the first portion is earned, then 8 clicks are required to earn each of the 5 points, and so on. The reinforcer not earned does not increase to the next level until it is earned. The testing session will end when participants no longer wish to earn points for access to either food choice. Water will be provided ad libitum. Participants are instructed on how to complete the computer task and will complete a practice session to demonstrate their understanding of the task. The task is completed with the experimenter in an adjacent room. Outcomes include the total number of responses (mouse-presses) performed for each type of food and the Pmax [29] of each choice, which is the last schedule that a participant met the response requirements for access to each food choice.

Physical activity reinforcement task. To assess the reinforcing value to be physically active, one computer station is set-up for the subject to earn access to physical activity (treadmill, elliptical ergometer, cycle ergometer) and the other computer station is set to earn access to sedentary alternatives (magazines, puzzles, card games). Access to the alternatives is dependent on earning points, which can be exchanged for the reinforcers using the schedules of reinforcement described above. For every 5 points earned, the subject will receive 5 min of access to exercise or 5 min of time to engage in the sedentary behavior, depending on the reinforcer that they were working for. Prior to the test participants will rate how much they like the exercise options and the sedentary alternative (APPENDIX 14) This sedentary alternative is provided to reduce the likelihood that participants would engage in responding for exercise out of boredom. This test will take place in the Human Performance Laboratory.

Body Composition. Body composition will be measured using a GE Lunar iDXA machine at the CCTS. A total body scan will be conducted with participants lying supine on the table and arms positioned to the side and palms flat on the table. Scans will be completed using the standard mode, unless the thick scan mode is suggested by the software. All scans will be analyzed using GE Lunar enCORE Software (13.60.033). Automatic edge detection will be used for scan analyses. The machine will be calibrated before each scanning session, using the GE Lunar calibration phantom. Outcomes will include total body lean mass, fat mass, bone mineral content and bone mineral density.

Each subject will undergo total body composition testing using a total body dual-energy x-ray absorptiometry (DXA) scan, and have their regional fat estimations performed using 3 circumference measures. Total body and regional, absolute and relative measures of soft tissue (fat, fat-free and mineral-free lean) masses will be made and analyzed by DXA scanning using a Lunar iDXA (GE Lunar Inc., Madison, WI; software version 13.10) using standardized procedures. The Lunar iDXA is the machine that is used during standard clinical testing. The waist, abdominal, and hip circumference measurements will be performed in triplicate using a flexible steel anthropometric tape (Rosscraft Anthrotape; Rosscraft Innovations Inc.) using standardized procedures. The body composition assessments testing will take place in the University of Kentucky Clinical Services Core (CSC) Functional Assessment and Body Composition Core (FAABC; inpatient suit 5th floor Chandler Medical Center) (CCTS).

Additional body composition tests will be performed on the Department of Dietetics and Human Nutrition's BodPod (air-displacement plethysmography) and the UK Athletics' DXA (Norland model) as a separate measure of internal reliability of these machines by comparing to the iDXA. The iDXA is the "gold standard" and will be used as the primary measure to test the current hypotheses.

Aerobic Fitness. A graded exercise treadmill test will be used to test aerobic fitness in addition to calculating rate of energy expenditure. Oxygen consumed and expired CO2 will be analyzed by indirect calorimetry. The test begins with a 5 minute warm-up of walking at 0% grade, 3.0 mph. Upon completion of the warm-up, the grade increases to 2.5% for 3 minutes with the speed fixed at 3.0 mph. The treadmill grade will then increase every 3 minutes to produce an approximately 10 beat/minute increase in heart rate from the previous stage. The test will continue until a heart rate of 85% HRR was attained or the participant fells they can no longer continue. The treadmill test will be performed at baseline, during week 6, and post training. The week 6 measurements will be used to adjust the intensity and duration of the exercise training sessions to account for improvements in aerobic fitness. Performance work capacity (PWC) will be utilized as a measurement of sub-maximal aerobic fitness with the rates of oxygen consumed at heart rates of 150 and 170 beats/minute serving as aerobic fitness outcomes.

Resting Metabolic Rate. Subjects will arrive to Funkhouser 117 fasted one morning prior to beginning the intervention (baseline) and 48 or more hours after their final exercise session of the intervention (week 13) to determine their RMR via indirect calorimetry (Cosmed USA, Chicago). This test lasts 45 minutes. Resting heart rate will be determined during the RMR test to be used to calculate HHR.

Hormone measurement. Subjects will report fasted to the CCTS and have an IV catheter placed to provide a fasted blood sample to analyze hormone and peptide concentrations associated with hunger and body weight regulation and complete VAS to determine hunger and satiety immediately prior to a standardized breakfast. The standardized breakfast will provide 20% of estimated energy needs for each individual based on their RMR and a sedentary activity factor of 1.4. Breakfast will consist of 2% milk and cornflakes (with the option of substituting unsweetened soy milk for those with a lactose sensitivity). Breakfasts will be consumed within 15 minutes. VAS scales for hunger and satiety and blood draws for hunger hormone measurement will be completed immediately before breakfast (-3hr) immediately after (-2.75), and every 15 minutes during the first hour (-2.5, -2.25, -2 hr) and then every 30 minutes thereafter (-1.5, -1, -0.5, 0) [30, 31]. Blood samples will be collected in EDTA-coated and serum tubes. Serum GLP-1, leptin, glucagon, and active grehlin will be measured using ELISA (Millipore, Phoenix Pharmaceuticals, Alpco). Serum insulin will be measured with a chemiluminescent immunometric assay (Siemens). Samples will be batch-analyzed to reduce interassay variability and stored at the CCTS until the conclusion of the study.

Habitual physical activity. For a 7 day period starting the day after subject's screening, 7 days following post-testing outcome assessments, and for 7 days during week 17, an ActiGraph accelerometer (GT3XPB model; Pensacola, Florida) will be worn to provide information regarding changes in habitual, free-living physical activity. Subjects will be instructed to wear it at the hip using the provided belt during all hours awake except when bathing or swimming. Data will be cleaned of non-wear time, defined as consecutive strings of zeros greater than 20 minutes. An epoch of 10 seconds will used for data collection. This will be used to measure weekly minutes of moderate to vigorous physical activity (MVPA) as well as minutes of sedentary activity and light intensity activity using the Crouter et.al algorithm [32], and Freedson cut-points [33].

Treatment Adherence. Subjects will be instructed to follow specific exercise plans that will elicit a 3,000 kcal energy expenditure per week. The length of the exercise session will depend on each individual's rate of energy expenditure. Each subject will be given a Polar heart rate monitor device to wear for each training session and meet with a research staff member weekly to download the previous week's exercise sessions to monitor compliance.

Tolerance for the discomfort of exercise. Discomfort tolerance will be measured by questionnaires. Subjects will complete the validated Preference for and Tolerance of the Intensity of Exercise Questionnaire (PRETIE-Q) at baseline and after training.

Energy and macronutrient intake. During weeks -3, 4, 8, 12, 17, participants will record their dietary intake for seven consecutive days.

Calculations. The accumulated energy balance (AEB) will be calculated from changes in FM and FFM as body composition changes reflect long-term alterations in energy balance (Rosenkilde et al. 13). Gains of 1kg FM or 1kg FFM will reflect 12,000 and 1,780 kcal, respectively (Elia et al., 2003). Losses of 1kg FM or 1kg FFM will be assumed to equal 9,417 and 884 kcal, respectively.

Exercise energy expenditure (ExEE) is calculated from the training-induced energy expenditure (TrEE) of 300 or 600 kcal/session with the addition of 15% excess post-exercise energy expenditure (Bahr, et al., 1997). The resting energy expenditure (REE) that would have occurred during the exercise sessions (REE x 1.2) will be subtracted. Thus, ExEE = (TrEE x 0.15) + (TrEE - training duration x REE 1.2).

The degree of compensation in response to the increase in ExEE is assessed through a compensation index calculated as (ExEE - AEB)/ExEE x 100%. When the compensation index equals zero AEB equals ExEE, or changes in body composition equal calories expended during exercise. Positive compensation suggests changes in body composition indicating a less negative energy balance than expected, whereas a larger than expected negative energy balance is referred to as negative compensation. Degree of compensation = (ExEE - AEB)/ExEE x 100%.

Statistical Analysis Plan: Baseline demographic and physical characteristics will be reported as means and standard errors. Baseline group (6 days/week, 2 days per week exercise, sedentary control) differences will be tested with one-way ANOVA. Alterations in accumulated negative energy balance, body composition, RRVfood, RRVexercise, dietary intake, energy expenditure, exercise discomfort, hunger/satiety hormones, and fitness will be tested with two-way repeated measures analysis of variance (RMANOVA) with group treated as a between-subjects variable and time treated as a within subjects variable. Power Analysis: The primary outcome is accumulated negative energy balance. Based on previous research the mean accumulated negative energy balances for 300 kcal of exercise and 600 kcal of exercise conditions were -83% + 100% (mean + SD) and 20% + 50%, respectively.

8. Resources:

The proposed study will utilize CCTS staff and facilities for measurement of hunger/satiety hormone concentrations, body composition (DEXA), and aerobic fitness tests. Laboratory space at Funkhouser includes a Quark RMR measurement equipment (Cosmed), NDS-R software for nutrition analysis, BodPod for air displacement plethysmography, and computers and space necessary for the food reinforcement task. The reinforcing value of exercise measurement will take place in the Human Performance Laboratory, where treadmills and cycle ergometers are available for participant use. The Department of Dietetics and Human Nutrition recently purchased new Polar A-300 heart rate monitors and ActiGraph accelerometers for the proposed study. Dr. Flack (PI) has led similar studies and may be training up to three graduate students that will assist in conducting the study.

9. Potential Risks:

DXA Scan. All subjects will be informed of the small amount of radiation they will receive while going through this procedure. Female subjects of childbearing potential will receive a urine pregnancy test prior to undergoing the DXA Scan. Those women found to be pregnant will not undergo the scan and will be removed from the study.

Blood Draw/ placement of IV catheter: Upon placement of the IV catheter, there may be some slight discomfort experienced from the insertion of the needle into the vein. Potential infection, soreness, pain, bleeding, bruising, and fainting may occur. This pain and soreness may last up to 24 hrs following the procedure. A trained nurse will place the IV catheter and standard precautions will be taken to guard against the following potential risks.

10. Safety Precautions:

Provisions to guard against the potential risks and discomforts discussed in section 9 are as follows: Every precaution to prevent a direct study injury will be taken by medical personnel and the investigators. Should an adverse or serious adverse event occur, the research participant will be followed by physicians, registered nurses and other research staff members for the duration of the participant's hospitalization. Routine care will be provided by the hospital staff. Emergency medical equipment, medications and supplies will be at the physician's disposal should the participants have an acute untoward reaction.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be overweight to obese (BMI 25-35 kg/m2) Not pregnant or lactating or planning to become pregnant in the next 6 months
* No limitations to safely participating in physical activity

Exclusion Criteria:

* Currently dieting to lose weight and no weight loss or gain >2kg over the past 3 months,
* Taking any medications that affect energy expenditure or eating,
* Regularly exercising (planned and structured aerobic or resistance activity).
* Participants must have no major health problems, cannot have known cardiovascular (cardiac, peripheral vascular, cerebrovascular), pulmonary (COPD, interstitial lung disease, cystic fibrosis) or metabolic (diabetes, thyroid disorders, renal or liver disease) disease.
* Tobacco use
* Have a medical condition that prevents safe exercise.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2019-08-18 (Actual); Study Completion 2019-08-18 (Actual)

PRIMARY OUTCOMES:
Accumulated Energy Balance | determined at 12 weeks by comparing to baseline data
  Change in energy balance assessed via DXA (weight loss)

SECONDARY OUTCOMES:
Compensation index | determined at 12 weeks by comparing to baseline data
  Degree of compensation for exercise-induced negative energy balance (energy expended - accumulated energy balance)/energy expended during exercise
Hormonal responses to meal and fasting levles | baseline to 12 weeks
  Changes in hunger hormone concentrations both fasting and in response to meal
Changes in dietary intake | baseline to 12 weeks
  Changes in dietary intake during the exercise intervention
Food reinforcment | baseline to 12 weeks
  Changes in food reinforcement after the exercise intervention
Exercise reinforcement | baseline to 12 weeks, 12 weeks to 16 weeks, baseline to 16 weeks.
  Changes in exercise reinforcement after the exercise intervention and after follow up
Habitual physical activity | baseline to 12 weeks, 12 weeks to 16 weeks, baseline to 16 weeks
  Changes in physical activity (accelerator counts)
Resting metabolic rate | baseline to 12 weeks
  Changes in resting metabolic rate after the exercise intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kyle D Flack, PhD, RD, Principal Investigator — University of Kentucky
Locations (1):
- Funkhouser Building, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Flack KD, Hays HM, Moreland J. Incentive sensitization for exercise reinforcement to increase exercise behaviors. J Health Psychol. 2021 Nov;26(13):2487-2504. doi: 10.1177/1359105320914073. Epub 2020 Apr 27. PMID 32338538